CLINICAL TRIAL: NCT00465478
Title: Autologous Bone Marrow Mononuclear Cell Transplantation in Treating Patients With Type 1 or 2 Diabetes Mellitus-a Phase 1/2 Study
Brief Title: Autologous Bone Marrow Mononuclear Cells Transplantation in Treating Diabetes Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL060308
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Bone Marros Mononuclear Cells; Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Autologous bone marrow mononuclear cell transplantation

SUMMARY:
The study evaluates the safety and efficiency of autologous bone marrow mononuclear cell transplantation in treating patients with type 1 or 2 Diabetes Mellitus. We hypothesize that autologous bone marrow stem cell transplantation will promote β-cells regeneration by directly differentiated from the transplanted BMMCs or stimulated local stem cells regeneration and thus decrease or eliminate the need of exogenous insulin and improve β-cells function.

DETAILED DESCRIPTION:
Patients with type 1 or 2 Diabetes mellitus will be recruited according to eligibility criteria. Bone marrow mononuclear cells (BMMCs) will be separated from the bone marrow aspirate of each patient and be directly delivered to pancreas via splenic artery with the distal lumen occlusion through an arterial catheter. All patients will be explained in details about the procedures involved in BMMC transplantation and sign the informed consent for the study; The Ethics Committee of Qilu hospital, ShanDong university approved the treatment protocol. All patients undergo scheduled follow-up evaluations for 5 years after transplantation. Clinical, hematological, metabolical evaluations are performed to analyses the effect of the transplant, Patients fitting the inclusion criteria but not agreeing to perform the transplantation are the control group and will received the regular OHA and/or insulin therapy .They are followed in parallel with transplanted patients and will be subjected to the same follow-up management including extensive endocrinological monitoring, diet and exercise program as transplantation patients during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes
* Between 16 to 65 years of age
* Requiring daily exogenous insulin injection for the glycaemic control
* With poor β-cell function
* Body mass index (BMI) < 28

Exclusion Criteria:

* Acute or chronic infections
* Chronic uncompensated organic insufficiency including heart, liver, renal and lung
* Any malignancies, congenital or acquired immunodeficiency
* Hematological diseases or coagulopathy
* Acute or chronic pancreatitis
* History of thoracic or abdominal aorta diseases
* Allergy to iodine
* Pregnancy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2006-03; Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Exogenous insulin requirement; Hemoglobin A1C; Glucose and C-peptide level;

SECONDARY OUTCOMES:
Safety assessment parameter: amylase, hepatic function,renal function,
lipid profile, autoantibody， Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Beihua Kong, MD PHD, Study Director — Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- See also: Related Info — http://www.qiluhospital.com